CLINICAL TRIAL: NCT03887286
Title: Feasibility and Accuracy of Focused Cardiac Ultrasound Using an FDA Approved Hand-held Ultrasound Device in Outpatient Setting in Our Institution.
Brief Title: Focused Cardiac Ultrasound
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Mary Sokoloski, Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20181089
Record Dates: First submitted 2019-03-21; First posted 2019-03-22 (Actual); Results first posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-05

CONDITIONS: Ventricular Dysfunction; Pericardial Effusion; Valvular Disease; Septal Defect
MeSH Terms: conditions — Ventricular Dysfunction; Pericardial Effusion; Heart Septal Defects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- treatment group (Experimental): All participants to receive standard transthoracic echocardiogram and hand held echocardiogram
  Interventions: Device: Philips EPIQ 7 ultrasound machine; Device: Philips Lumify Broadband sector array transducer

INTERVENTIONS:
Device: Philips EPIQ 7 ultrasound machine — Standard transthoracic echocardiography
Device: Philips Lumify Broadband sector array transducer — Portable hand-held ultrasound device

SUMMARY:
To compare the images from standard cardiac ultrasound with images from a small hand-held device; to find out more about the feasibility and accuracy of a small hand-held ultrasound device.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to pediatric cardiology clinic at Holtz Children's hospital requiring comprehensive or limited transthoracic echocardiogram.
* Willing and able to provide informed consent or assent.
* In clinically stable condition as assessed by the principal investigator..
* With adequate echocardiographic windows.

Exclusion Criteria:

* Patients with poor echocardiographic windows.
* Patients who refuse informed consent.
* Pregnant women.
* Prisoners.
* Patients deemed unfit to participate in the clinical trial as assessed by the principal investigator.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Sokoloski, M.D., Principal Investigator — University of Miami
Locations (1):
- Jackson Memorial Hospital, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Group
Started | 47
Completed | 47
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Group
Number analyzed (Participants) | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.8 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
weight [Mean (Standard Deviation); unit: kg] | 27.24 (23.41)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Detected With Ventricular Dysfunction, Pericardial Effusion, Valvular Disorders, Septal Disorders, and Coronary Anomalies.
Description: Comparison of diagnostic ability of portable hand-held cardiac ultrasound with standard transthoracic echocardiography
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Groups:
- Standard Transthoracic Echocardiogram Intervention: The transthoracic echocardiogram was performed and read via Intersocietal Commission Accreditation Echocardiography Laboratories (ICAEL) standard
- Hand Held Echocardiography: The hand held echocardiogram was performed and read via Intersocietal Commission Accreditation Echocardiography Laboratories (ICAEL) standard
Arm/Group | Standard Transthoracic Echocardiogram Intervention | Hand Held Echocardiography
Number analyzed (Participants) | 47 | 47
Participants
  normal anatomy | 13 | 13
  minor cardiac abnormality | 9 | 4
  major cardiac abnormality | 25 | 23

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/47
Serious Adverse Events (participants affected / at risk) | 0/47
Other Adverse Events (participants affected / at risk) | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2018-12-17): https://cdn.clinicaltrials.gov/large-docs/86/NCT03887286/Prot_000.pdf